CLINICAL TRIAL: NCT04153903
Title: Integrated Coronary Multicenter Imaging Registry - Extended
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0476
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with intermediate lesions: Imaging cohort will be performed invasive angiography and optical coherence tomography (or Coronary CT angiography) with FFR(Fractional Flow Reserve) values of the intermediate lesions (50-70% stenosis)
  Interventions: Other: OCT, coronary angiography, FFR

INTERVENTIONS:
Other: OCT, coronary angiography, FFR — Coronary images by OCT and angiography and FFR values will be registered.

SUMMARY:
The coronary images of invasive angiography and optical coherence tomography (or Coronary CT angiography) with FFR(Fractional Flow Reserve) values of the intermediate lesions (50-70% stenosis) will be prospectively registered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent coronary CT angiography because of chest pain
2. Patients who need OCT or FFR evaluation because of intermediate lesions according to invasive angiography (diameter stenosis of 50-70%)
3. Age: 20-80 yrs
4. Patients who consent and fully understand the protocol
5. Patients who consent the clinical follow-up
6. Patients who can be followed-up

Exclusion Criteria:

1. Patients who had contrast allergy
2. Patients who had unstable blood pressure needing the vasopressors
3. Patients who had severe left ventricular function (left ventricular ejection fraction<30%)
4. Chronic kidney disease who had Cr level of greater than 2.0 mg/dl
5. Patients whose expected survival is less than 12 months
6. Patients who had a severe valvular disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of computed FFR derived by coronary images and real FFR values | at registration
  FFR values computed by OCT/CT/invasive coronary angiography will be compared by real invasive FFR values

SECONDARY OUTCOMES:
Adverse event (Death, acute myocardial infarction) | 2 years after registration
  Death and occurrence of myocardial infarction during follow-up period will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Cardiovascular Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No